CLINICAL TRIAL: NCT06213142
Title: Developing the Unified Protocol-Single Session Experience Platform for Adolescent Mental Health
Acronym: CBToolkit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3-C Institute for Social Development (Industry)
Collaborators: University of Miami (Other); Stony Brook University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3CG078
Record Dates: First submitted 2023-12-29; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Depression; Depression, Anxiety; Depression in Adolescence; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants in the acceptability test will be assigned to the same set of study tasks, where all participants will engage with the two modules and provide feedback. All participants will complete the RCADS pre and post, in addition to all study-related surveys: demographics, pre- and post-knowledge checks, module component ratings, prototype evaluations, and advocacy ratings. All participants will be invited to the follow-up focus group sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBToolkit (Experimental): CBToolkit includes two SSI modules: (1) Mindful Awareness, with the goal of increasing awareness and tolerance of physical sensations and emotional experiences using mindfulness practices and tips and (2) Flexible Problem Solving, with the goal of promoting cognitive flexibility, applying problem-solving strategies in difficult scenarios, and learning to modify behavioral action tendencies.
  Interventions: Other: CBToolkit

INTERVENTIONS:
Other: CBToolkit — CB Toolkit Mindful Awareness module to increase awareness and tolerance of physical sensations and emotional experiences using mindfulness practices. The module involves videos with motion graphics, video demos, voiceover, music, and sound effects intermixed throughout with a variety of interactive exercises tailored to specific core components. The module aims to establish understanding of the intervention concept (psychoeducation), increase self-efficacy in mindfulness skills via active practice and personalized feedback, and facilitate self-reflection and understanding of strengths and improvement areas related to mindfulness. CBToolkit Flexible Problem Solving module to promote cognitive flexibility, applying problem-solving strategies in difficult scenarios, and learning to modify behavioral action tendencies. Videos and activities will be tailored to provide examples of effective problem-solving techniques and provide personalized reinforcing and/or scaffolded feedback.

SUMMARY:
This SBIR Phase I proposal will develop and test the acceptability and feasibility of a new suite of digital Single-Session Interventions, specifically applying Unified Protocol core principles for emotional disorders, to produce a highly accessible, engaging, and scalable product to help address the clinical needs of youth.

DETAILED DESCRIPTION:
This project proposes develop a suite of Single Session Intervention (SSI) modules using the Unified Protocol (UP) core principles. For Phase I, the team will develop two SSI modules from UP: Awareness of Physical Sensations and Emotional Experiences, and Being Flexible in Your Problem Solving. For the acceptability test (Specific Aim 2), investigators will recruit 60 youth who are screened as eligible based on the internalizing subscale of the Pediatric Symptom Checklist. Caregivers/parents of youth will be recruited using targeted social media advertisements, where they can view a brief study description and complete the eligibility screener. If interested, caregivers can provide contact information for the study team to conduct consent and assent processes. Following consent and enrollment, participants will receive private login information to access the prototype and study materials. First, participants will complete pre-surveys that collect demographic information and responses to the Revised Children's Anxiety and Depression Scale (RCADS). Next, participants will take a brief survey to assess knowledge of intervention concepts presented in the first module: Mindful Awareness. Then, they will engage with the module and provide feedback on the quality of its components. Then, they will complete the knowledge assessment again. Participants will complete the same process for the second module: Flexible Problem Solving (pre knowledge check, review, rate the quality, and post knowledge check). Participants will complete a product evaluation to rate their overall experience with the prototype (quality, usability, innovation, feasibility, and value) and the degree they advocate for full product development. Finally, participants will take the RCADS at the end of the review period. There will also be an opportunity for participants to participate in a brief feedback call to provide additional feedback.

ELIGIBILITY:
Inclusion Criteria:

* be ages 13 to 17 years old
* be willing and available to take part in the study requirements
* be fluent in English
* have access to the internet with a mobile device or personal computer
* have parent permission
* screen as eligible according to the internalizing subscale from the Pediatric Symptom Checklist

Exclusion Criteria:

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Program Feedback Scale for Adolescents | 2 week followup post module review
  Adolescents will complete this 12-item measure, rating the extent to which they agree with statements about the usability, acceptability, and feasibility of the CBToolkit modules. The measure includes 9 Likert items and 3 open-ended items. Responses to the Likert items range from 1 (Really Disagree) to 5 (Really Agree). Total scores are based on the Likert items are range from 0 to 45. Higher scores reflect more positive opinions.
Module Knowledge | Average of 2 weeks apart, as pre- and post-tests
  Adolescents will complete this 9-item measure to determine what they know about key concepts taught in the CBToolkit module prior to and following review of the modules. The measure includes 9 multiple choice items with a 1 correct response per item. Total scores are based on the number of items with correct responses and range from 0 to 9. Higher scores reflect more correct responses.
Revised Children's Anxiety and Depression Scale- Shortened | Average of 2 weeks apart, as pre- and post-tests
  Adolescents will complete the shortened 11-item version of this measure to assess levels of anxiety and depression prior to and following review of the modules. The measure includes 11 Likert items. Responses to the Likert items range from 0- Never to 3- Always. Total scores are based on the Likert items are range from 0 to 33. Higher scores reflect more severe symptoms.

SECONDARY OUTCOMES:
Usage Metrics from the CBToolkit system for adolescents | The period in which adolescents interact with the system, approximately 2 weeks
  The CBToolkit software will tracks progress through the modules, and the length of time spent on each sections of the module. These metrics are measured in seconds. A longer time generally indicates more time spent with the content.
Feedback interviews with adolescents | 15-minutes, completed after the test of the CBToolkit system
  Adolescents will participate in individual interviews. They will be asked about their experience with the CBToolkit, strengths and weaknesses of CBToolkit, and challenges to using CBToolkit.. Comments will be combined and grouped based on themes in a qualitative summary.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa DeRosier, PhD, Principal Investigator — 3C Institute; Jill Ehrenreich-May, PhD, Principal Investigator — University of Miami; Jessica Schleider, PhD, Principal Investigator — StoneyBrook University
Locations (1):
- 3C Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No